CLINICAL TRIAL: NCT05565677
Title: Prognostic Value of Lung Cancer MicroAnatomy in Three Dimensions: a Micro-CT Based Trial
Brief Title: Prognostic Value of Lung Cancer MicroAnatomy in 3D
Acronym: LungCaMa3D
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: National and Kapodistrian University of Athens (Other); University of Southampton (Other)
Responsible Party: Principal Investigator, Dimitrios Moysidis, Principal Investigator, Aristotle University Of Thessaloniki
Other Study IDs: 5039
Record Dates: First submitted 2022-09-29; First posted 2022-10-04 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Lung Cancer; Adenocarcinoma of Lung; Pathology; Micro-computed Tomography; X-ray Histology; Digital Pathology
Keywords: micro-CT; lung cancer; digital pathology
MeSH Terms: conditions — Lung Neoplasms; Adenocarcinoma of Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Lung tissue specimens will be surgically resected according to clinical indications (per standard of care) in patients with presumptive clinical diagnosis of lung cancer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patients with lung cancer: Patients with a presumptive diagnosis of lung cancer for whom surgical resection or sampling will be clinically indicated according to the standard practices of the Cardiothoracic Department of AHEPA University Hospital of Thessaloniki, will be enrolled in this prospective study once they give written informed consent for specimen imaging. Surgical resections will be performed per standard of care and there will be no difference in patients' clinical management depending on the acquisition or not of surgical specimens. Patients with altered mental status and those who are unable or unwilling to provide informed consent will be excluded from this study.
  Interventions: Device: micro-computed tomography scanning of lung tissue specimens

INTERVENTIONS:
Device: micro-computed tomography scanning of lung tissue specimens — Micro-computed tomography will be utilized to scan surgically resected lung tissue specimens.

SUMMARY:
Micro-computed tomography (micro-CT) is a novel biomedical non-destructive, slide-free digital imaging modality, which enables the rapid acquisition of accurate high-resolution, volumetric images of intact surgical tissue specimens. This imaging modality provides microscopic level of detail of intact tissues in three-dimensions without requiring any specimen preparation. Its non-destructive nature and the ongoing enhancement of imaging resolution and contrast renders micro-CT imaging particularly well suited for microanatomic studies in basic research across a wide range of interventional medical disciplines, including oncology.

Our proposal concerns a multidisciplinary basic research effort which aims to facilitate the effective identification of different -and maybe challenging to differentiate- lung cancer patterns based on 3D X-ray histology. As an alternative for the use of hematoxylin & eosin (H&E) slides, optimized micro-CT scanning of soft tissues emerges as a promising tool to enable non-invasive 3D X-ray histology of formalin-fixed and paraffin-embedded (FFPE) lung cancer specimens.

The objective of our proposal is to offer novel insights into the complex architecture of each lung cancer subtype after imaging FFPE surgical specimens, resected from lung cancer surgeries. The investigators aim to generate 3D datasets of FFPE lung cancer tissues which will be combined with the corresponding conventional 2D histology slides. Our study will be also adequately empowered to identify particular differences in morphometric measurements according to each particular lung cancer growth pattern.

Finally, this proposal aims to delineate the different 3D microanatomy and morphology of some patterns that are challenging to interpret and differentiate through traditional 2D histological evaluation, such as papillary and lepidic adenocarcinoma growth patterns.

Classification of the histological subtypes based on 2D histology sections can be ambiguous, as shown by suboptimal inter-observer consensus when determining predominant histological subtypes in FFPE lung adenocarcinoma tissue specimens. Hence, micro-CT-based 3D imaging of the lung specimens could aid classification of histological subtypes by providing more comprehensive sampling of the entire tissue block and yielding detail relevant for subtype classification that might not be visible in 2D sections alone.

DETAILED DESCRIPTION:
Patients with a presumptive diagnosis of lung cancer for whom surgical resection or sampling will be clinically indicated according to the standard practices of the Cardiothoracic Department of AHEPA University Hospital of Thessaloniki, will be enrolled in this prospective study once they give written informed consent for specimen imaging. Surgical resections will be performed per standard of care and there will be no difference in patients' clinical management depending on the acquisition or not of surgical specimens. Patients with altered mental status and those who are unable or unwilling to provide informed consent will be excluded from this study.

Sample preparation Following surgical resection, human lung tissue specimens will be placed in a sterile container by the surgeon in the operating room. Choice of container will be based on specimen size. Right after the end of the operation, each specimen will be fixed in neutral buffered formalin for 48 hours in tissue cassettes and will be embedded in paraffin wax following a standardized protocol.

Imaging protocol After the collection of the formalin-fixed and paraffin-embedded (FFPE) surgically resected lung cancer specimens, these will be transported to the μ-VIS X-ray Imaging Centre at the University of Southampton in accordance with particular biological material transfer agreement. The FFPE lung samples will be scanned at the μ-VIS X-ray Imaging Centre using a custom-built Nikon Metrology micro-CT scanner according to standardized protocol.

Histological assessment Following non-destructive micro-CT imaging, the scanned FFPE specimens will be transported to the Pathology Laboratory of the First Pathology Department of the National and Kapodistrian University of Athens in accordance with particular biological material transfer agreement. The specimens will be set in paraffin blocks for sectioning. After sectioning, sections will be de-paraffinized and stained using Movat's pentachrome stain. The sections will be imaged and assessed histologically by an experienced and "blinded" pulmonary pathologist (S.T.). The pathologist will also assess a number of non-scanned FFPE lung cancer specimens to confirm the non-destructive nature of micro-CT imaging for the resected specimens. Identification of radiation-induced or ischemic alterations, deviant necrosis or cellular degeneration could be indicative outcomes of a destructive imaging method.

Statistical analysis The generated imaging data will be statistically analyzed using Bland-Altman plots to determine intra- and inter-observer variability in the interpretation of micro-CT imaging data. Wilcoxon's rank sum test or Kruskal Wallis's test will be utilized to evaluate any differences within specific morphometric measurements (percent object volume, object surface/volume ratio, object surface density, structure model index, structure thickness, structure linear density, structure separation, connectivity, connectivity density) among different growth patterns. All statistical analyses will be performed with SPSS (version 27) and a p-value of less than 0.05 will be considered as the threshold of statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a presumptive diagnosis of lung cancer for whom surgical resection or sampling will be clinically indicated.

Exclusion Criteria:

* Patients with altered mental status and those who are unable or unwilling to provide informed consent for specimen imaging.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a presumptive diagnosis of lung cancer for whom surgical resection or sampling will be clinically indicated according to the standard practices of the Cardiothoracic Department of AHEPA University Hospital of Thessaloniki, will be enrolled in this prospective study once they give written informed consent for specimen imaging. Surgical resections will be performed per standard of care and there will be no difference in patients' clinical management depending on the acquisition or not of surgical specimens. Patients with altered mental status and those who are unable or unwilling to provide informed consent will be excluded from this study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between micro-CT and histopathological findings | 2 years
  After co-registration of micro-CT and histopathological images via relevant software (e.g., ImageJ plugin: UnwarpJ elastic registration), a blinded pathologist (S.T.) will assess the co-aligned images to assess whether the investigator can identify the presence of lung cancer based on the generated 3D micro-CT images. The outcomes of this qualitative analysis will be statistically analyzed using Bland-Altman plots to determine intra- and inter-observer variability in the interpretation of micro-CT imaging data.
Evaluation of specific morphometric measurements according to lung cancer type | 2 years
  Wilcoxon's rank sum test or Kruskal Wallis's test will be utilized to evaluate any differences within specific morphometric micro-CT based measurements among different growth patterns. All statistical analyses will be performed with SPSS (version 27) and a p-value of less than 0.05 will be considered as the threshold of statistical significance.

IPD SHARING:
Plan to Share IPD: No